CLINICAL TRIAL: NCT01459783
Title: Comparative Effectiveness of Dementia Care Strategies in Underserved Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Olive View-UCLA Education & Research Institute (Other); Alzheimer's Association (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HQ217RC4; 1RC4AG038804-01 (NIH)
Record Dates: First submitted 2011-01-18; First posted 2011-10-26 (Estimated); Results first posted 2015-05-22 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Dementia
Keywords: Caregivers; Comparative Effectiveness Research; Cost Effectiveness; Patient Care Management; Social Work
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dementia care management in person (Active Comparator): The dementia care management protocol will be delivered via face-to-face interactions in participants' homes or in mutually convenient locations between a trained care manager and the care recipient/informal family caregiver dyad, supplemented by telephone.
  Interventions: Behavioral: Dementia care management
- Dementia care management telephone only (Active Comparator): The dementia care management protocol will be delivered via telephonic meetings only. Assessment, education, counseling, and social support procedures as well as referral and follow-ups will follow the same procedural content as stipulated for the face-to-face intervention, however, contact will not be planned in person.
  Interventions: Behavioral: Dementia care management

INTERVENTIONS:
Behavioral: Dementia care management — Care management is initiated via a structured assessment, to identify prevalent caregiving problems: unmet need for assistance, lack of social support, educational needs, difficulty with managing behavioral issues and safety concerns, need for respite, establishing advance care planning, depression of the person with dementia as well as the caregiver, management of other chronic medical issues, and need for diagnostic information and assistance with acute medical issues. Collaboration between the caregiver and the care manager results in problem prioritization and subsequent counseling, education, referrals as needed, and proactive follow-up to achieve resolution of these problems. An electronic tracking tool and resource manual guide delivery of the care management protocols.

SUMMARY:
Dementia is a condition that is growing in prevalence and which harms not only the afflicted individual but also adversely affects the health of their family and other informal caregivers. New methods for delivering comprehensive assistance to persons with dementia and their caregivers are known to be effective and can delay nursing home placement, but this study will discover 1) whether more face-to-face involvement rather than telephone delivery of this assistance will work better among poor patients in Los Angeles, and 2) if one method is better than the other, what are the differences in costs between them. These data will enable administrators in public health care settings around the US and non-profit foundations addressing dementia patient and caregiver needs to decide what method provides the best value and the best outcome relative to its cost.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers of persons with dementia
* Caregivers must either live with the care recipient (person with dementia) or be the identified primary support
* Caregiver relationship must have been present for the prior 6 months
* Caregivers must have telephone access
* Caregivers must speak English or Spanish
* Care recipients must have a prior dementia diagnosis
* Care recipients must be living in the community other than a nursing facility

Exclusion Criteria:

* Persons with dementia, lacking an informal caregiver who can communicate in Spanish or English, or living in a long term care facility
* Caregiver lacks the capacity to consent to study participation

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2011-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Chodosh, M.D., MSHS, Principal Investigator — RAND; Barbara Vickrey, M.D., MPH, Principal Investigator — RAND
Locations (1):
- Olive View-UCLA Medical Center, Sylmar, California, United States

REFERENCES:
- [Result] Chodosh J, Colaiaco BA, Connor KI, Cope DW, Liu H, Ganz DA, Richman MJ, Cherry DL, Blank JM, Carbone Rdel P, Wolf SM, Vickrey BG. Dementia Care Management in an Underserved Community: The Comparative Effectiveness of Two Different Approaches. J Aging Health. 2015 Aug;27(5):864-93. doi: 10.1177/0898264315569454. Epub 2015 Feb 4. PMID 25656074

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult caregivers (CG) lived with dementia care recipient (CR) or were the main support for >6 months. CRs had to live in the community (no nursing home). Admin data (ICD-9 codes) yielded eligible CRs from Olive View Med Center+local clinics. CRs got recruitment mailings to give to CG. CG were also recruited at CR's memory clinic+community outreach
Pre-assignment Details: A research assistant (RA) got informed consent either in-person at clinic or by phone for outreach/admin data sources. Contact info was sent to the survey group who completed enrollment and a baseline survey; then participants were randomized by the RA. Between the survey and randomization, 3 CGs were found ineligible and 4 duplicates were found.
Groups:
- Dementia Care Management in Person: The dementia care management protocol will be delivered via face-to-face interactions in participants' homes or in mutually convenient locations between a trained care manager and the care recipient/informal family caregiver dyad, supplemented by telephone.
  Dementia care management: Care management is initiated via a structured assessment, to identify prevalent caregiving problems: unmet need for assistance, lack of social support, educational needs, difficulty with managing behavioral issues and safety concerns, need for respite, establishing advance care planning, depression of the person with dementia as well as the caregiver, management of other chronic medical issues, and need for diagnostic information and assistance with acute medical issues. Collaboration between the caregiver and the care manager results in problem prioritization and subsequent counseling, education, referrals as needed, and proactive follow-up to achieve resolution of these problems.
- Dementia Care Management Telephone Only: The dementia care management protocol will be delivered via telephonic meetings only. Assessment, education, counseling, and social support procedures as well as referral and follow-ups will follow the same procedural content as stipulated for the face-to-face intervention, however, contact will not be planned in person.
  Dementia care management: Care management is initiated via a structured assessment, to identify prevalent caregiving problems: unmet need for assistance, lack of social support, educational needs, difficulty with managing behavioral issues and safety concerns, need for respite, establishing advance care planning, depression of the person with dementia as well as the caregiver, management of other chronic medical issues, and need for diagnostic information and assistance with acute medical issues. Collaboration between the caregiver and the care manager results in problem prioritization and subsequent counseling, education, referrals and proactive follow-up.
Period: Baseline to 6 Months
Arm/Group | Dementia Care Management in Person | Dementia Care Management Telephone Only
Started | 71 | 73
Completed | 39 | 53
Not Completed | 32 | 20
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 12 | 6
Not completed — Lost to Follow-up | 19 | 14
Period: 6 Months to 12 Months
Arm/Group | Dementia Care Management in Person | Dementia Care Management Telephone Only
Started | 39 | 53
Completed | 20 | 23
Not Completed | 19 | 30
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Lost to Follow-up | 2 | 7
Not completed — Study ended before 12-month follow-up | 11 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dementia Care Management in Person | Dementia Care Management Telephone Only | Total
Number analyzed (Participants) | 71 | 73 | 144
Age, Continuous [Mean (Standard Deviation); unit: years] — This is the caregiver age.
  years | 48.07 (14.28) | 50.95 (12.71) | 49.53 (13.53)
Sex: Female, Male [Count of Participants; unit: Participants] — This is the caregiver's gender
  Participants
    Female | 48 | 46 | 94
    Male | 23 | 27 | 50
Race/Ethnicity, Customized [Number; unit: participants] — This is the caregiver's race/ethnicity
  participants
    African American | 6 | 3 | 9
    Caucasian or Euro-American | 7 | 6 | 13
    Hispanic or Latino | 52 | 60 | 112
    Other | 6 | 4 | 10
Education [Number; unit: participants] — This is the caregiver's educational attainment
  participants
    Less than high school | 25 | 27 | 52
    High school graduate or GED | 19 | 13 | 32
    Some college or 2-year degree | 12 | 22 | 34
    4-year college or more | 15 | 11 | 26
Language spoken with friends and family [Number; unit: participants] — This is the caregiver's language spoken with friends and family
  participants
    English | 25 | 24 | 49
    Spanish | 39 | 46 | 85
    Other | 7 | 3 | 10
Relationship type to care recipient [Number; unit: participants] — This is the caregiver's relationship to the care recipient/person with dementia.
  participants
    Spouse | 9 | 16 | 25
    Son/Daughter | 36 | 41 | 77
    Brother/sister | 1 | 1 | 2
    Cousin/other relative | 6 | 1 | 7
    Other | 19 | 14 | 33

OUTCOME MEASURES:

1. Primary Outcome: Change in Caregiver Burden at 6 and 12 Months
Description: The Zarit Burden Interview (BI) is a widely used validated measure to assess stressors experienced by caregivers of persons with dementia. Originally a 29-item instrument, the 22-item modified version is easily completed by telephone. This instrument covers five constructs of burden: health, psychological well-being, finances, social life, and relationship with impaired person and an overall summary score of caregiver burden. Higher Zarit scores indicate greater caregiver burden. The minimum possible score is 0, and the maximum possible score is 110.
Time Frame: 0, 6 and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dementia Care Management in Person | Dementia Care Management Telephone Only
Number analyzed (Participants) | 71 | 73
units on a scale
  Unadjusted score at 6 months | 29.99 (17.51) | 30.09 (19.6)
  Unadjusted score at 12 months | 28.1 (18.53) | 28.13 (11.84)
  Baseline score | 30.07 (16.99) | 30.91 (17.98)
Statistical Analysis 1: Comparison: Dementia Care Management in Person vs Dementia Care Management Telephone Only; Analyses were intention-to-treat. Due to attrition and those ineligible for 12-month follow-up due to study ending before that time, we created survey non-response weights for each wave. Prior to the study, a sample size of 125 participants per group was based on the two primary outcomes, with a Type I Error of 0.025 (Bonferroni adjustment), setting a 0.5-SD difference in outcomes as clinically important, 80% power, 0.45 SD difference in difference in outcomes between groups, and 25% attrition; Test type: Superiority or Other; p = 0.76, Regression, Linear — We adopted Bonferroni adjustment for multiple testing and used a significance level of .05/3 = 0.017 to interpret the results for our primary outcomes; Multivariate analyses included non-response weights and controlled for study arm, stratification variables, baseline values, & intervention duration; Mean Difference (Final Values) = 0.91, 95% CI 2-sided [-5.13 to 6.95] — The difference in differences at 12 months is reported as in-person arm minus phone arm values from a multivariable analysis. A positive adjusted difference means worse burden for the in-person arm compared to the phone arm

2. Primary Outcome: Change in Care Recipient Memory and Problem Behaviors at 6 and 12 Months
Description: The Revised Memory and Behavior Problem Checklist (RMBPC) was developed by Teri and colleagues. The RMBPC instrument assess 24 care receiver problems in the areas of behavior, memory, and depression and whether each behavior had occurred in the prior week. Higher RMBPC scores mean worse memory/behavior problems. The minimum possible score for number of problems is zero, and the maximum score for number of problems is 24.
Time Frame: 0, 6 and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dementia Care Management in Person | Dementia Care Management Telephone Only
Number analyzed (Participants) | 71 | 73
units on a scale
  unadjusted 6 month post intervention | 9.68 (5.53) | 8.53 (5.33)
  12 month unadjusted post-intervention | 8.2 (5.86) | 9.26 (5.26)
  Baseline score | 9.44 (4.92) | 9.43 (5.27)
Statistical Analysis 1: Comparison: Dementia Care Management in Person vs Dementia Care Management Telephone Only; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.49, Regression, Linear — We used Bonferroni adjustment for multiple testing and a significance level of .05/3 = 0.017 to interpret the results for our primary outcomes. The behavior measure is analyzed two ways: total number of problems (reported here), and reaction score; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-1.74 to 3.55] — The difference in differences at 12 months is reported as in-person arm minus phone arm values from a multivariable analysis. A positive adjusted difference means worse problems for the in-person arm compared to the phone arm

3. Secondary Outcome: Change in Caregiver Depression at 6 and 12 Months
Description: The Patient Health Questionnaire - Nine (PHQ-9) is a 9-item self-report measure of depressive symptoms over the previous 2 weeks. The PHQ-9 is the depression module of the PRIME- MD diagnostic instrument for common mental disorders. It covers each of the 9 DSM-IV depression criteria scoring them as "0" (not at all) to "3" (nearly every day).
Time Frame: 0, 6 and 12 months
Reporting Status: Not Posted

4. Secondary Outcome: Change in Caregiver Quality of Life at 6 and 12 Months
Description: The Caregiver-Targeted Quality of Life (CG-QOL) measure covers 10 dimensions of QOL relevant to caregivers of persons with dementia, incorporates non-health related issues as well as positive aspects of caregiving, and has demonstrated feasibility as a phone-based instrument in both English and Spanish. Eighty items are distributed across 10 scales: assistance with ADLs, assistance with IADLs, personal time, role limitation due to caregiving, family involvement, demands of caregiving, worry, caregiver feelings, spirituality and faith, benefits of caregiving.
Time Frame: 0, 6 and 12 months
Reporting Status: Not Posted

5. Secondary Outcome: Change in Care Recipient Quality of Life at 6 and 12 Months
Description: The investigators will evaluate patient health-related quality of life (HRQOL) by proxy (caregiver) assessment using the 15-item Health Utilities Index (HUI2), a generic health state classification system with preference-based utility weights derived from the general population. The HUI is one of the more widely used utility measures and has been used in previous studies of elderly with dementia and their caregivers.
Time Frame: 0, 6 and 12 months
Reporting Status: Not Posted

6. Secondary Outcome: Change in Process Measures of Dementia Care Quality at 6 and 12 Months
Description: The investigators will collect caregiver survey identified care process measures to assess which medical care processes that are specific to dementia occurred as a potential mediator of change in outcomes.
Time Frame: 0, 6 and 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Dementia Care Management in Person | Dementia Care Management Telephone Only
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/73
Other Adverse Events (participants affected / at risk) | 0/71 | 0/73

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No